CLINICAL TRIAL: NCT04799899
Title: Mindfulness-Based Cognitive Therapy Delivered Via Group Videoconferencing for Acute Coronary Syndrome Patients With Depressive Symptoms: A Pilot RCT
Brief Title: MBCT Via Group Videoconferencing for Acute Coronary Syndrome Patients With Depressive Symptoms: A Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christina Luberto, Assistant Professor, Department of Psychiatry, Harvard Medical School; Staff Psychologist, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000544
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome; Depression
Keywords: Mindfulness; Acute Coronary Syndrome; Videoconferencing; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual MBCT Intervention (Experimental): Participants will participate in 8 weekly virtual group sessions of MBCT. Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30-60 minutes).
  Interventions: Behavioral: Adapted MBCT
- Virtual Health Enhancement Control (Experimental): Participants will participate in 8 weekly virtual group sessions that focus on cardiac health and depression education. Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30-60 minutes).
  Interventions: Behavioral: Cardiac Health Enhancement

INTERVENTIONS:
Behavioral: Adapted MBCT — The adapted MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health.
  Arms: Virtual MBCT Intervention
Behavioral: Cardiac Health Enhancement — The cardiac health enhancement control group will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will learn about depression and cardiac health.
  Arms: Virtual Health Enhancement Control

SUMMARY:
The aim of this study is to establish, in a pilot RCT (approx. N=50 participants) with a time- and attention-matched health enhancement control, (a) the feasibility of the recruitment procedures (screening, eligibility, enrollment rates), and feasibility and acceptability of the (b) MBCT and control interventions (adherence, retention, fidelity, satisfaction, group videoconferencing delivery) and (c) data collection procedures by group (adherence, satisfaction). Hypothesis 1a: Recruitment will be feasible as evidenced by screening, eligibility, and enrollment rates; (1b) the MBCT and control interventions and (1c) data collection procedures in both groups will be feasible and acceptable.

DETAILED DESCRIPTION:
The current study will employ an open pilot RCT with a time-and-attention-matched health control group to determine the feasibility and acceptability of a virtual, MBCT intervention for ACS patients. The investigators plan to enroll approximately N=50 participants (approx. 3 MBCT groups and approx. 3 health enhancement control groups with approximately 6-7 participants per group; accounting for 20% attrition). Participants will be randomized to a MBCT or a time- and attention-matched health enhancement control in a 1:1 design using a random number generator. Participants will then be stratified by antidepressant medication use. The MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health. The health enhancement control group will follow the same structure of the MBCT intervention (e.g., 8 virtually-delivered MBCT sessions, approximately 1.5 hours each) and will educate participants on depression and cardiac health (e.g., relationship between depression and cardiac health, cardiac risk factors, cardiac health behaviors, finding resources for mental health care). Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30-60 minutes).

Participants will be recruited through EPIC, the hospital's clinical data registry, advertisements (e.g., flyers, brochures) placed throughout the hospital, direct provider referrals, and from inpatient cardiac units. Patients who express interest in the study will be asked complete an eligibility screening. Eligible patients agreeable with study participation will then complete informed consent with study staff prior to enrollment.

Participants will be enrolled in either one of three MBCT intervention cohorts (approx.) or one of three health enhancement control cohorts (approx.). Participants in all of these groups will be expected to participate in 8-weekly, 1.5-hour virtual sessions. Participants in the MBCT intervention group will be expected to participate in 30 minutes of at-home daily practice. Participants in the health enhancement control group will be expected to review educational videos or readings between sessions. A licensed mental health provider (e.g., LICSW, PhD) trained in the MBCT protocol will delivered the intervention to the MBCT intervention group. A licensed clinician or pre-doctoral or post-doctoral fellow with supervision from a licensed clinician will lead the control group. Both the MBCT intervention and health enhancement control groups will be delivered via Zoom, secure, HIPPA-compliant video-conferencing software.

Study assessments will include a battery of self-report surveys administered at baseline, post-intervention, and 3-month follow-up; session satisfaction surveys administered after each intervention session; post-intervention individual exit interviews (conducted via telephone or videoconference); blood spot samples self-collected by participants at baseline, post-intervention, and 3-month follow-up (submitted to the research team via paper mail); and, for the MBCT-intervention group, home practice logs submitted between each intervention session. Primary outcomes for the intervention are feasibility and acceptability. Exploratory outcomes are changes in emotional and biological variables. Data collected from this study will generate knowledge about e-health technologies and congruent research methods to apply to other mind-body interventions and patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Lifetime ACS per medical record and/or patient confirmation
2. Current elevated depression symptoms (PHQ-9 greater than or equal to 5)
3. Age 35-85 years
4. Access to high-speed internet

Exclusion Criteria:

1. Active suicidal ideation or past-year psychiatric hospitalization (per patient report and/or medical record review)
2. Non-English-speaking
3. Cognitive impairments preventing informed consent per medical record review and/or cognitive Screen less than or equal to 4
4. Patient deemed unable to complete the study protocol or has a condition that would likely interfere with the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Luberto, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mongan Institute: Health Policy Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tully PJ, Ang SY, Lee EJ, Bendig E, Bauereiss N, Bengel J, Baumeister H. Psychological and pharmacological interventions for depression in patients with coronary artery disease. Cochrane Database Syst Rev. 2021 Dec 15;12(12):CD008012. doi: 10.1002/14651858.CD008012.pub4. PMID 34910821

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 407 participants recruited, 219 were screened. 63 were found ineligible and 108 declined to participate leaving 48 eligible participants. 18 refused to participate so 30 participants were consented to the study. 6 of those 30 consented participants did not complete the baseline survey or withdrew from the study, leaving 24 participants to be randomized into the intervention groups.
Period: Overall Study
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Started | 12 | 12
Completed | 10 (Defined by: completion of post intervention survey) | 8 (defined by: completion of post intervention survey)
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the baseline survey and were randomized into a study arm.
Groups:
- Virtual Mindfulness Based Cognitive Therapy (MBCT) Intervention: Participants will participate in 8 weekly virtual group sessions of MBCT. Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30-60 minutes).
  Adapted MBCT: The adapted MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health.
- Total: Total of all reporting groups
Arm/Group | Virtual Mindfulness Based Cognitive Therapy (MBCT) Intervention | Virtual Health Enhancement Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.92 (10.950) | 57.42 (12.266) | 57.67 (11.374)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: score on scale] — The Patient Health Questionnaire-9 (PHQ-9) was used to assess depression. There are 9 items in this scale and the minimum score is 0 and maximum score is 27. Higher scores indicate higher severity of depression.
  score on scale | 9.67 (4.097) | 12.42 (6.543) | 11.04 (5.521)
Time Since Acute Coronary Syndrome (ACS) [Mean (Standard Deviation); unit: Years] | 3.38 (3.844) | 2.39 (1.77) | 2.88 (2.97)
Type of Acute Coronary Syndrome (ACS) [Count of Participants; unit: Participants]
  Myocardial infarction (MI) | 1 | 0 | 1
  Non-ST-elevation myocardial infarction (NSTEMI) | 3 | 5 | 8
  Spontaneous coronary artery dissection (SCAD) | 3 | 3 | 6
  Unstable Angina (UA) | 1 | 0 | 1
  ST-elevation myocardial infarction (STEMI) | 2 | 0 | 2
  SCAD & NSTEMI | 0 | 1 | 1
  NSTEMI & STEMI | 1 | 0 | 1
  SCAD & STEMI | 0 | 1 | 1
  MI & STEMI | 0 | 1 | 1
  NSTEMI & UA & SCAD | 0 | 1 | 1
  STEMI & UA | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility: Percent of Participants Screened Eligible
Description: Feasibility outcomes for recruitment will include: >70% meet screening criteria
Time Frame: 6 months
Population: The number of participants who were screened.
Measure: Count of Participants; unit: Participants
Groups:
- Screened Participants: This group contains all participants who were screened as part of the study enrollment process.
Arm/Group | Screened Participants
Number analyzed (Participants) | 219
Participants | 48

2. Primary Outcome: Recruitment Feasibility: Percent of Participants Enrolled
Description: Feasibility outcomes for recruitment will include: >70% of eligible enroll
Time Frame: 6 months
Population: Participants who were deemed eligible in the study screening process.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: This group contains all participants who were deemed eligible in the study screening process.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 48
Participants | 24

3. Primary Outcome: MBCT Feasibility: Percent of Participants Retained
Description: MBCT intervention feasibility will include: >75% of participants retained at post-assessment survey
Time Frame: 6 months
Population: MBCT feasibility outcome only; Control Group was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 12
Participants | 10

4. Primary Outcome: Mindfulness Based Cognitive Therapy (MBCT) Feasibility: Percent of Participants Adherent to Treatment
Description: MBCT intervention feasibility will include: >75% of participants attending 6/8 sessions. "Adherent to treatment" is defined as participants attending 6 out of 8 sessions.
Time Frame: 6 months
Population: MBCT outcome measure only; control group was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 12
Participants | 6

5. Primary Outcome: Mindfulness Based Cognitive Therapy (MBCT) Feasibility: Percent of Participants Adherent to Home Practice
Description: MBCT feasibility will include: >75% complete home practice at least 3 days/week. Adherence was defined as completion of home practice long at least 3 days per week.
Time Frame: 6 months
Population: Participants (n = 10) in the MBCT intervention who completed the post intervention survey. Control group was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 10
Participants | 8

6. Primary Outcome: Control Group Feasibility: Percent of Participants Retained
Description: Control group feasibility will include: >75% of participants retained at post-assessment survey
Time Frame: 6 months
Population: MBCT intervention group was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 12
Participants | 8

7. Primary Outcome: Control Group Feasibility: Percent of Participants Adherent to Treatment
Description: Control group feasibility will include: >75% of participants attending 6/8 sessions sessions. "Adherent to treatment" is defined as participants attending 6 out of 8 sessions.
Time Frame: 6 months
Population: MBCT Intervention Group was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 12
Participants | 8

8. Primary Outcome: Control Group Feasibility: Percent of Participants Adherent to Home Practice
Description: Control group feasibility will include: >75% complete home practice at least 3 days/week. "Adherent to home practice" is defined as participants completing home practice at least 3 days per week.
Time Frame: 6 months
Population: N = 8 participants completed the post intervention survey. MCBT intervention group was not analyzed for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 8
Participants | 4

9. Primary Outcome: Videoconferencing Feasibility: Number of Sessions Missed Due to Technical Problems
Description: Videoconferencing feasibility will be assessed by: <20% of sessions missed due to technical problems
Time Frame: 6 months
Population: All participants who were randomized into study groups. Across all groups/arm, there were 32 sessions in the study.
Measure: Count of Units; unit: Videoconferencing sessions
Units Other Than Participants: Videoconferencing sessions
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Number analyzed (Participants) | 12 | 12
Number analyzed (Videoconferencing sessions) | 16 | 16
Videoconferencing sessions | 0 | 0

10. Primary Outcome: Blood Spot Feasibility: Percent of Blood Spot Samples Submitted at Baseline
Description: Blood spot feasibility will be assessed by >75% of samples submitted at baseline. Participants contributed one blood spot sample at the specified time point.
Time Frame: At Baseline (Month 0)
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Number analyzed (Participants) | 12 | 12
Participants | 11 | 11

11. Primary Outcome: Blood Spot Feasibility: Percent of Blood Spot Samples Submitted at Post-intervention
Description: Blood spot feasibility will be assessed by >75% of samples submitted at post-intervention
Time Frame: At Post Intervention (Month 3)
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Virtual Health Enhancement Group: Participants will participate in 8 weekly virtual group sessions of MBCT. Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30-60 minutes).
  Adapted MBCT: The adapted MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health.
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Group
Number analyzed (Participants) | 12 | 12
Participants | 8 | 7

12. Primary Outcome: Mindfulness Based Cognitive Therapy (MBCT) Acceptability: Ratings of Intervention Satisfaction
Description: MBCT acceptability will be assessed by overall program satisfaction (1=not at all, 10=very much). Satisfaction will be measured by mean score greater than 7.5
Time Frame: At post intervention (Month 3)
Population: Participants who answered intervention satisfaction question on post intervention survey. Control Group was not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 9
score on a scale | 8.67 (2.598)

13. Primary Outcome: Mindfulness Based Cognitive Therapy (MBCT) Acceptability: Percent of Participants Who Plan to Continue Using the Skills
Description: MBCT and acceptability will be assessed by 75% plan to use the skills
Time Frame: 6 months
Population: Participants who answered the relevant survey question on the post intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 8
Participants | 8

14. Primary Outcome: Mindfulness Based Cognitive Therapy (MBCT) Acceptability: Percent of Participants Who Would Recommend the Program
Description: MBCT and acceptability will be assessed by >75% of participants reporting that they would recommend the program to others
Time Frame: 6 months
Population: Number of participants who answered the relevant survey question on the post intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT Intervention
Number analyzed (Participants) | 8
Participants | 8

15. Primary Outcome: Control Group Acceptability: Ratings of Intervention Satisfaction
Description: Control group acceptability will be assessed by overall program satisfaction (1=not at all, 10=very much). Satisfaction will be measured by an overall mean score greater than 7.5.
Time Frame: 6 months
Population: Number of participants who answered the relevant survey question on the post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 8
score on a scale | 8.13 (1.959)

16. Primary Outcome: Control Group Acceptability: Percent of Participants Who Plan to Continue Using the Skills
Description: Control group acceptability will be assessed by 75% of participants reporting that they plan to use the skills
Time Frame: 6 months
Population: Number of participants who answered the relevant survey question on the post-intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 8
Participants | 8

17. Primary Outcome: Control Group Acceptability: Percent of Participants Who Would Recommend the Program
Description: Control group acceptability will be assessed by >75% of participants reporting that they would recommend the program to others
Time Frame: 6 months
Population: Number of participants who answered the relevant survey question on the post-intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Health Enhancement Control
Number analyzed (Participants) | 8
Participants | 8

18. Primary Outcome: Videoconferencing Acceptability: Ratings of Videoconferencing Satisfaction
Description: Videoconferencing acceptability will be assessed in terms of overall satisfaction (1=poor,10=excellent; M>7.5)
Time Frame: 6 months
Population: Participants who answered intervention satisfaction questions on post intervention survey.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Number analyzed (Participants) | 8 | 8
Units on a scale | 9.75 (.463) | 9.63 (1.061)

19. Primary Outcome: Blood Spot Acceptability: Blood Spot Collection Ease
Description: Blood spot acceptability will be assessed by ratings of ease of data collection (1=not at all, 10=extremely). Satisfaction will be measured by an overall mean score greater than 7.5.
Time Frame: 6 months
Population: Participants who answered videoconferencing satisfaction question on post intervention survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Number analyzed (Participants) | 10 | 8
units on a scale | 8.50 (2.121) | 8.38 (3.159)

20. Primary Outcome: Blood Spot Acceptability: Blood Spot Collection Comfort
Description: Blood spot acceptability will be assessed by ratings of ease of level of pain (1=very much pain, 10=very little pain; M>8.0). Acceptability will be measured by an overall mean score greater than 8.0.
Time Frame: 6 months
Population: Participants who answered videoconferencing satisfaction question on post intervention survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
Number analyzed (Participants) | 10 | 8
units on a scale | 9.10 (1.595) | 9.50 (1.069)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Virtual MBCT Intervention | Virtual Health Enhancement Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04799899/Prot_SAP_000.pdf